CLINICAL TRIAL: NCT07203391
Title: TRIUMPH - Tebentafusp and Roginolisib in Uveal Melanoma to Prolong T-cell Homeostasis
Brief Title: Tebentafusp and Roginolisib in Uveal Melanoma to Prolong T-cell Homeostasis
Acronym: TRIUMPH
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Professor, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIUMPH
Record Dates: First submitted 2025-09-21; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Uveal Melanoma, Metastatic
Keywords: tebentafusp; Roginolisib
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Standard Tebentafusp with the addition of Roginlisib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination (Experimental): Tebentafusp/ Roginolisib
  Interventions: Drug: roginolisib

INTERVENTIONS:
Drug: roginolisib — Investigational combination - initially at 40mg (Dose 1) then 80mg (Dose 2)

SUMMARY:
This is a combination study of Tebentafusp and the PI3Kdelta inhibitor, Roginolisib

DETAILED DESCRIPTION:
Based on the established activity of Tebentafusp, and the promising action of Roginolisib, this trial combines the two drugs from cycle 4 onwards in patients with metastatic uveal melanoma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants must be aged 18 years or over at the time, to be eligible to participate in this study.
2. Histologically or cytologically confirmed metastatic UM or unresectable UM patients
3. HLA-A*02:01 positive
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
5. Currently undergoing first-line treatment for mUM with tebentafusp
6. Tebentafusp related toxicity, including cytokine release syndrome that has resolved to grade ≤ 1 as per CTCAE v5.0.
7. Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control (eg double barrier) from the trial screening date until 6 months after the final dose of the program intervention; cessation of birth control after this point shall be discussed with a responsible physician.
8. Pregnant or lactating women are prohibited from enrolling on this program.
9. Male participants are not allowed to donate sperm from the time of enrolment until 6 months post- administration of program interventions.

Exclusion Criteria:

1. Presence of untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or cord compression. NOTE: Participants with treated CNS lesions may enroll provided all of the following apply:

   1. Treated CNS lesions must be radiographically stable for ≥ 4 weeks after intervention (surgery and/or radiation).
   2. Participants must be neurologically stable off systemic corticosteroids for at least 2 weeks prior to trial entry
2. Ongoing Grade 2 or greater treatment related toxicity due to tebentafusp
3. Prior treatment with a PI3Kδ inhibitor
4. Prior Grade 4 cytokine release syndrome related to Tebentafusp
5. Systemic treatment with steroids or any other immunosuppressive drug use within 2 weeks of the planned first dose of program intervention, with the following exceptions:

   1. Treatment for well-controlled and asymptomatic adrenal insufficiency is permitted, but replacement dosing is limited to prednisone ≤ 10 mg daily or the equivalent.
   2. Local or topical steroid therapies (eg, optic, ophthalmic, intra- articular, or inhaled medications) are acceptable.
   3. Premedication for allergy to contrast reagent.
6. Any relevant medical condition, which in the opinion of the treating physician, would prevent the participant enrolling into the Program due to concerns related to safety, compliance with procedures, or interpretation of program results.
7. Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications.
8. Chronic viral infections as indicated below. NOTE: Testing for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) status prior to enrollment is not necessary unless clinically indicated.
9. Known HIV infection unless all of the following are applicable:

   1. Receiving an approved, stable, effective combination antiretroviral therapy regimen for ≥3 months prior to the planned first study intervention
   2. CD4 T-cell count >350 cells/µl
   3. CD4 T-cell nadir (lowest historical count) < 350 cells/µl
   4. Viral load confirmed as <50 copies/ml during Screening.
10. Known HBV infection, unless on stable anti-viral therapy for > 4 weeks prior to the planned first dose of program intervention and viral load confirmed as undetectable during Screening.
11. Known HCV infection, unless the participant has received curative treatment, and viral load was confirmed as undetectable during Screening.
12. Participant with an out-of-range Screening laboratory values defined as shown below. NOTE: Hematology evaluations must be performed ≥ 7 days from any blood or blood product transfusion and ≥ 14 days from any dose of hematologic growth factor.

    1. Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 30 mL/minute.
    2. Total bilirubin > 1.5 × ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin > 1.5 × ULN.
    3. Alanine aminotransferase > 5 × ULN in the presence of liver metastases; > 3 X ULN if not
    4. Aspartate aminotransferase > 5 × ULN in the presence of liver metastases ; > 3 X ULN if not
    5. Platelet count < 75 × 109/L
    6. Hemoglobin < 9 g/dL
13. Clinically significant cardiac disease or impaired cardiac function, including any of the following:

    1. Congestive heart failure (New York Heart Association Class ≥ 3)
    2. QTcF>470msec at baseline
    3. Uncontrolled hypertension defined as systolic blood pressure [BP] > 160 mmHg or diastolic BP > 110 mmHg with the following requirements:
    4. If initial measurement is elevated, additional assessments should be taken where each assessment is the mean value of 3 measurements taken at least 5 minutes apart.
    5. Eligibility is based on the average of at least 2 assessments taken at least 1 hour apart.
    6. Acute myocardial infarction or unstable angina pectoris < 6 months prior to the planned first dose of program intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
• To determine the safety and tolerability of roginolisib and tebentafusp in HLA-A*02:01 positive patients advanced uveal melanoma (UM). | Through study completion, estimated average of 1 year
  CTCAE V5.0
• To establish a maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of the combination of roginolisib and tebentafusp in HLA-A*02:01 positive patients advanced uveal melanoma (UM). | Through study completion, estimated average of 1 year
  As determined by DSMB

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, MBBS PhD FRACP, Principal Investigator — St Vinents Hospital sydney
Locations (2):
- Australia (2):
  - St Vincents Hospital, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Confidentiality